CLINICAL TRIAL: NCT02198807
Title: A Phase IIa Proof of Concept Study to Explore the Efficacy, Tolerability and Safety of Fosmidomycin Sodium When Administered With Piperaquine Tetraphosphate to Adults and Older Children With Acute Uncomplicated Plasmodium Falciparum Malaria
Brief Title: Evaluation of Fosmidomycin and Piperaquine in the Treatment of Acute Falciparum Malaria
Acronym: FOSPIP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jomaa Pharma GmbH (Industry)
Collaborators: Centre de Recherche Médicale de Lambaréné (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JP017
Record Dates: First submitted 2014-07-22; First posted 2014-07-24 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Oral Treatment of Acute Uncomplicated Plasmodium Falciparum Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fosmidomycin-Piperaquine (Experimental): Fosmidomycin sodium capsules 450 mg, dosage: 30mg/kg twice daily for 3 days Piperaquine phosphate tablets 320 mg, dosage: 16 mg/kg once a day for 3 days
  Interventions: Drug: Fosmidomycin-Piperaquine

INTERVENTIONS:
Drug: Fosmidomycin-Piperaquine

SUMMARY:
The objective of this study is to explore the role of fosmidomycin and piperaquine as non-artemisinin-based combination therapy for acute uncomplicated Plasmodium falciparum when administered over three days.

Together, fosmidomycin and piperaquine fulfil the WHO criteria for combination therapy by meeting the three key parameters of having different modes of action and different biochemical targets while exhibiting independent blood schizonticidal activity. Like the artemisinins, fosmidomycin is fast-acting, has an excellent safety record and is active against existing drug-resistant parasites. Piperaquine has a long half life protecting fosmidomycin as a much shorter lived molecule against selection of resistant parasites and will provide post-treatment prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 1 to 60 years inclusive
* Body weight between 5kg and 90kg inclusive
* Acute manifestations of a mono-infection with Plasmodium falciparum as determined by either a rapid diagnostic test for adults or microscopically confirmed by an asexual parasitaemia of 1,000 to 150,000/uL and fever with an axillary temperature of > 37.5 degress C or oral/rectal/tympanic temperature of > 38.0 degrees C or history of fever during the previous 72 hours
* Compliance with contraceptive measures throughout the study period of 63 days in females of child bearing potential

Exclusion Criteria:

To be eligible for inclusion in the study, subjects must NOT meet any of the following criteria:

* Signs of severe/complicated malaria according to WHO criteria
* Pregnancy as excluded by negative serum human chorionic gonadotrophin (hCG) test
* Lactation
* Mixed Plasmodium infection
* Severe vomiting on three or more occasions in the previous 24 hours
* Severe diarrhoea on four or more occasions in the previous 24 hours
* Concomitant disease masking assessment of response including

  * abnormal liver function tests with bilirubin > 40 µmol/L, aspartate aminotransferase (ASAT) and alanine aminotransferase (ALAT) levels > x 2 upper limit of normal
  * impaired renal function with creatinine level > x 2 upper limit of normal
  * haemoglobin level < 7.5g/dl
  * white cell count > 12000/µL
* History of cardiovascular disease including arrhythmia with QTc interval ≥ 450msec, respiratory disease including active tuberculosis, hepatic disease including jaundice, renal failure, malignancy, neurological disorders including convulsions and psychiatric disturbances
* History of immunological disease including Hepatitis A, B and C and HIV-AIDS
* Severe malnutrition
* History of hypersensitivity or adverse reactions to fosmidomycin, piperaquine, artesunate and mefloquine
* Treatment with antimalarial and antibacterial agents within the previous 28 days

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Per protocol, PCR-corrected cure rate on Day 28 | 28 days
  Six-hourly asexual counts until negative on three successive occasions.
  Weekly smears on days 7, 14, 21 and 28

SECONDARY OUTCOMES:
Per protocol, PCR-corrected cure rates on Day 7 and Day 63 | 63 days
  Weekly smears on days 35 +/- 3 days, 42 +/- 3 days and 63 +/- 3 days
Derived parasite reduction ratio at 48 hours | 2 days
  Six-hourly asexual counts until negative on three successive occasions
Parasite clearance time | 96 hours
  Six-hourly asexual counts until negative on three successive occasions
Fever clearance time | 96 hours
  Six hourly temperature recordings until normal on three successisve occasions
Proportion of subjects with gametocytes on Day 7 | 7 days
  Smear on Day 7
Adverse event recording | 28 days
  Recording of vital signs and ECG monitoring
  Recording of incidence, severity, drug-relatedness and seriousness of AEs and laboratory abnormalites

REFERENCES:
- [Derived] Mombo-Ngoma G, Remppis J, Sievers M, Zoleko Manego R, Endamne L, Kabwende L, Veletzky L, Nguyen TT, Groger M, Lotsch F, Mischlinger J, Flohr L, Kim J, Cattaneo C, Hutchinson D, Duparc S, Moehrle J, Velavan TP, Lell B, Ramharter M, Adegnika AA, Mordmuller B, Kremsner PG. Efficacy and Safety of Fosmidomycin-Piperaquine as Nonartemisinin-Based Combination Therapy for Uncomplicated Falciparum Malaria: A Single-Arm, Age De-escalation Proof-of-Concept Study in Gabon. Clin Infect Dis. 2018 Jun 1;66(12):1823-1830. doi: 10.1093/cid/cix1122. PMID 29293893